CLINICAL TRIAL: NCT04308512
Title: A Comprehensive Care Coordination and Management Platform for Alzheimer's Disease and Related Dementia (Care4AD)
Brief Title: Care Coordination System for People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bijan Najafi, PhD (Other)
Collaborators: BioSensics (Industry)
Responsible Party: Sponsor-Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-46087
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease; Dementia; Dementia Alzheimers
Keywords: Alzheimber; Dementia; care coordination
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group: Care coordination with active Nili System (Active Comparator): Participants in the intervention group will receive the Active Nili system. Essential activities of daily living (ADL) were pre-programmed by a care coordination expert for the Active Nili Care Phase. In addition, patients and their caregivers were able to schedule supplementary tasks through the Nili App. All feedback features were fully activated in the Active Nili device.
  Interventions: Behavioral: Active Nili device
- Control Group: Receiving passive Nili device (Active Comparator): Participants in the control group will receive the passive Nili device with preprogrammed care coordination and limited daily programming. However, all reminders and activity of daily living (ADL) task scheduling will remain deactivated during this phase.
  Interventions: Behavioral: Passive Nili system

INTERVENTIONS:
Behavioral: Active Nili device — Eligible dyads, consisting of individuals with dementia (IWD) and their caregivers, will be randomized in a 1:1 ratio to receive either a 3-month Passive Nili Care device or a 3-month Active Nili Care device. Both devices are identical in design and feature a kiosk-mode interactive tablet that supports IWD in following preprogrammed daily routines, including instrumental activities of daily living (IADLs), social engagement, phone calls, photo sharing, medication adherence, and listening to music or audiobooks. In the Active Nili device, all reminders and programming features will be enabled, whereas in the Passive device, these functions will remain disabled. In both groups, essential ADL tasks will be preprogrammed by a care coordination expert. In addition, the Active Nili system will allow patients and caregivers to schedule personalized tasks through the Nili app.
  Arms: Intervention Group: Care coordination with active Nili System
Behavioral: Passive Nili system — Eligible dyads, consisting of individuals with dementia (IWD) and their caregivers, will be randomized in a 1:1 ratio to receive either a 3-month Passive Nili Care device or a 3-month Active Nili Care device. Both devices are identical in design and feature a kiosk-mode interactive tablet that supports IWD in following preprogrammed daily routines, including instrumental activities of daily living (IADLs), social engagement, phone calls, photo sharing, medication adherence, and listening to music or audiobooks. In the Active Nili device, all reminders and programming features will be enabled, whereas in the Passive device, these functions will remain disabled. In both groups, essential ADL tasks will be preprogrammed by a care coordination expert. In addition, the Active Nili system will allow patients and caregivers to schedule personalized tasks through the Nili app.
  Arms: Control Group: Receiving passive Nili device

SUMMARY:
Dementia, a chronic disease of aging, is characterized by progressive cognitive decline that interferes with independent functioning. The medical, psychological, social and functional sequelae of dementia cause great stress to patients, their caregivers, and their family. The investigator proposes to examine effectiveness of a home-based care coordination and management device, called Care4AD (Nili device) to help caregivers effectively coordinate, manage, and improve dementia care.

DETAILED DESCRIPTION:
In this study, the investigator will evaluate the effectiveness of a supportive care coordination device, Care4AD/Nili, in reducing caregiver burden and stress, improving adherence to scheduled tasks, and increasing engagement among individuals with dementia (IWD).

A 3-month randomized controlled trial (RCT) will be conducted with an anticipated 100 caregiver-patient dyads, consisting of 50 individuals with dementia or cognitive impairment and their 50 primary caregivers. Dyads will be randomized in a 1:1 ratio to receive either (1) a Passive Nili device (preprogrammed care coordination with limited daily programmability) for three months, or (2) an Active Nili device for three months. The Active Nili device offers interactive, personalized programming with real-time notifications, task logging, and enhanced social and cognitive engagement features, including photo sharing, phone calls, music, and audiobooks.

The primary outcome is change in caregiver burden. Secondary outcomes include usability metrics such as perceived ease of use, perceived benefit, technology-related anxiety, and overall attitudes toward adoption.

ELIGIBILITY:
Inclusion Criteria include:

* Caregivers (>18 years old) taking care of older patients (> 55 years old) with mild or moderate Alzheimer's Disease or self-reported memory problems and MOCA score of 26 or lower.
* Must be ambulatory
* Must be in a residential home with a caregiver/informant.

Exclusion Criteria:

* Immobility or inability to engage in activities that are essential for independent living (e.g., patients with severe dementia);
* Any significant medical or psychiatric condition that, in the judgment of the investigators, would potentially interfere with the ability to participate in the study
* Major hearing/visual impairment;
* Residing in a nursing home or are receiving hospice care;
* Inability to communicate in English or Spanish;
* Unavailability or unwillingness of the caregiver of the patient to attend the interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mishra RK, Park C, Momin AS, Rafaei NE, Kunik M, York MK, Najafi B. Care4AD: A Technology-Driven Platform for Care Coordination and Management: Acceptability Study in Dementia. Gerontology. 2023;69(2):227-238. doi: 10.1159/000526219. Epub 2022 Sep 12. PMID 36096091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible dyads will consist of individuals with dementia (IWD) and their caregivers. For this study, outcomes related to caregivers will be presented, as the primary endpoint is the reduction of caregiver burden.
Groups:
- Intervention Group: Care coordination with active Nili System: Participants in the intervention group received the Active Nili system. Essential activities of daily living (ADL) were pre-programmed by a care coordination expert for the Active Nili Care Phase. In addition, patients and their caregivers were able to schedule supplementary tasks through the Nili App. All feedback features were fully activated in the Active Nili device.
Period: Overall Study
Arm/Group | Intervention Group: Care coordination with active Nili System | Control Group: Receiving passive Nili device
Started | 28 (The numbers reported in the Participant Flow Milestones represent the number of dyads (individuals with dementia or cognitive impairment and their caregivers). However, the primary outcome is reported only for caregivers, as the focus of this study is on reducing caregiver burden.) | 38 (The numbers reported in the Participant Flow Milestones represent the number of dyads (individuals with dementia or cognitive impairment and their caregivers). However, the primary outcome is reported only for caregivers, as the focus of this study is on reducing caregiver burden.)
Number of caregivers | 14 | 19
Number of patients | 14 | 19
Completed (A total of 54 participants completed the study, including 22 (11 caregiver-patient dyads) in the intervention group and 32 (16 caregiver-patient dyads) in the control group) | 22 | 32
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Population: A total of 66 participants were recruited, including 28 (14 caregiver-patient dyads) in the intervention group and 38 (19 caregiver-patient dyads) in the control group
Groups:
- Intervention Group: Care coordination with active Nili System: Dyad participants in the intervention group received the Active Nili system. Essential activities of daily living (ADLs) were preprogrammed by a care coordination expert, and patients and their caregivers could schedule additional tasks through the Nili App. All feedback features were fully activated during the Active Nili Care phase.
  The demographics and caregiver outcomes are presented in this report.
- Control Group: Care coordination with passive Nili System: Dyad participants in the control group will receive the passive Nili device with preprogrammed care coordination and limited daily programming. However, all reminders and activity of daily living (ADL) task scheduling will remain deactivated during this phase.
  The demographics and caregiver outcomes are presented in this report.
- Total: Total of all reporting groups
Arm/Group | Intervention Group: Care coordination with active Nili System | Control Group: Care coordination with passive Nili System | Total
Number analyzed (Participants) | 28 | 38 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: A total of 66 participants were recruited, including 28 (14 caregiver-patient dyads) in the intervention group and 38 (19 caregiver-patient dyads) in the control group
  years
    Caregivers: number analyzed (Participants) | 14 | 19 | 33
    Caregivers | 63.4 (13.5) | 53 (17.3) | 57.7 (16.3)
    Patients: number analyzed (Participants) | 14 | 19 | 33
    Patients | 70.8 (13.4) | 70.0 (11.0) | 70.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 66 participants were recruited, including 28 (14 caregiver-patient dyads) in the intervention group and 38 (19 caregiver-patient dyads) in the control group
  Participants
    Caregivers: number analyzed (Participants) | 14 | 19 | 33
    Caregivers: Female | 10 | 14 | 24
    Caregivers: Male | 4 | 5 | 9
    Patients: number analyzed (Participants) | 14 | 19 | 33
    Patients: Female | 9 | 9 | 18
    Patients: Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 66 participants were recruited, including 28 (14 caregiver-patient dyads) in the intervention group and 38 (19 caregiver-patient dyads) in the control group
  Participants
    Caregivers: number analyzed (Participants) | 14 | 19 | 33
    Caregivers: Hispanic or Latino | 0 | 2 | 2
    Caregivers: Not Hispanic or Latino | 2 | 15 | 17
    Caregivers: Unknown or Not Reported | 12 | 2 | 14
    Patients: number analyzed (Participants) | 14 | 19 | 33
    Patients: Hispanic or Latino | 3 | 2 | 5
    Patients: Not Hispanic or Latino | 9 | 16 | 25
    Patients: Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 66 participants were recruited, including 28 (14 caregiver-patient dyads) in the intervention group and 38 (19 caregiver-patient dyads) in the control group
  Participants
    Caregivers: number analyzed (Participants) | 14 | 19 | 33
    Caregivers: American Indian or Alaska Native | 0 | 0 | 0
    Caregivers: Asian | 1 | 1 | 2
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 9 | 9 | 18
    Caregivers: White | 3 | 6 | 9
    Caregivers: More than one race | 1 | 1 | 2
    Caregivers: Unknown or Not Reported | 0 | 2 | 2
    Patients: number analyzed (Participants) | 14 | 19 | 33
    Patients: American Indian or Alaska Native | 0 | 0 | 0
    Patients: Asian | 1 | 1 | 2
    Patients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Patients: Black or African American | 7 | 9 | 16
    Patients: White | 3 | 6 | 9
    Patients: More than one race | 1 | 1 | 2
    Patients: Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Burden and Stress of Caregivers Over 3 Months
Description: Caregiver burden and stress will be assessed using the 12-item short version of the Zarit Burden Interview (ZBI), a validated survey for dementia caregivers. The ZBI evaluates caregivers' experiences across emotional, physical, and social domains, capturing the strains and difficulties associated with their role. Items address issues such as perceived decline in personal health, the impact of caregiving on relationships with family and friends, and overall feelings of burden. Percentage change from baseline to 3 months will be calculated. Change from baseline burden was reported only for caregivers.
  Percentage change on the ZBI-12 can range from -100% (complete resolution of burden) to a large positive increase, with negative values indicating improvement and positive values indicating worsening; reductions of 20% or more are generally considered clinically meaningful improvements.
Time Frame: Baseline, 3 months
Population: Change from baseline burden was reported only for caregivers.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Intervention Group: Care coordination with active Nili System | Control Group: Receiving passive Nili device
Number analyzed (Participants) | 11 | 16
percentage change | -52.0 (61.9) | -31.9 (101.3)

2. Secondary Outcome: Acceptability, Perception of Benefit, and Ease of Use of Care4AD
Description: This will be assessed using technology acceptance model (TAM) survey adopted for telehealth applications
Time Frame: 3 months
Reporting Status: Not Posted, anticipated posting 2025-10

3. Secondary Outcome: Change in Baseline Quality of Life at 3 Months: Global PROMIS-10
Description: Quality of life will be assessed using a validated questionnaire, called Global PROMIS-10.
  The adult PROMIS Global Health measure produces two scores: Physical Health and Mental Health. The "7+2" scales include the same global health score plus one fatigue and one pain interference item which are scored independently.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Number of Adverse Events Over 3 Month Study
Description: Adverse events, including falls, dehydration, urinary tract infections, and emergency department visits, were systematically monitored over a 3-month period. These events were reported exclusively for patients.
Time Frame: During the 3 month study
Population: Adverse events were reported for patients.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: Care coordination with active Nili System: Participants in the control group received active Nili system. Essential activity daily living (ADL) tasks will be pre-programmed by our care coordination expert for the Active Nili Care Phase. Patients and their caregivers in the intervention group will be also able to schedule additional tasks.
  Active Nili device: Eligible dyads, consisting of individuals with dementia (IWD) and their caregivers, will be randomized in a 1:1 ratio to receive either a 3-month Passive Nili Care device or a 3-month Active Nili Care device. Both devices are identical in design and feature a kiosk-mode interactive tablet that supports IWD in following preprogrammed daily routines, including instrumental activities of daily living (IADLs), social engagement, phone calls, photo sharing, medication adherence, and listening to music or audiobooks. In the Active Nili device, all reminders and programming features will be enabled, whereas in the Passive device, these functions will remain disabled. In both groups, essential ADL tasks will be preprogrammed by a care coordination expert. In addition, the Active Nili system will allow patients and caregivers to schedule personalized tasks through the Nili app.
Arm/Group | Intervention Group: Care coordination with active Nili System | Control Group: Receiving passive Nili device
Number analyzed (Participants) | 14 | 19
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Intervention Group: Care coordination with active Nili System: Dyad participants in the intervention group received the Active Nili system. Essential activities of daily living (ADL) were pre-programmed by a care coordination expert for the Active Nili Care Phase. In addition, patients and their caregivers were able to schedule supplementary tasks through the Nili App. All feedback features were fully activated in the Active Nili device.
- Control Group: Receiving passive Nili device: Dyad participants in the control group will receive the passive Nili device with preprogrammed care coordination and limited daily programming. However, all reminders and activity of daily living (ADL) task scheduling will remain deactivated during this phase.
Arm/Group | Intervention Group: Care coordination with active Nili System | Control Group: Receiving passive Nili device
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/19
Other Adverse Events (participants affected / at risk) | 0/14 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT04308512/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT04308512/ICF_001.pdf